CLINICAL TRIAL: NCT04366882
Title: Increasing Our Understanding of COVID-19: Minimal Invasive Autopsies to Investigate Clinical, Radiological, Microbiological and Histopathological Changes in Deceased COVID-19 Patients
Brief Title: Minimal Invasive Autopsies to Investigate Changes in Deceased COVID-19 Patients
Acronym: MIA-COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jessa Hospital (Other)
Collaborators: Hasselt University (Other); University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: JessaH_COVID-19_MIA
Record Dates: First submitted 2020-04-22; First posted 2020-04-29 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: COVID-19; cause of death; pathophysiology
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CT-scan with minimal invasive autopsy — CT-guided biopsies will be performed directly following the diagnostic CT-scan. Biopsies will be taken from heart, liver, lungs, spleen, kidneys and abdominal fat according to a standard operation procedure. Biopsies will be taken for further histological examination and storage in the biobank. Of the lung, additional samples will be taken for microbiological examination. Additional samples will be taken in case of (focal) abnormalities on CT-imaging. In case of pleural, cardiac or abdominal fluid, this will be aspirated for further cytological, biochemical and microbiological examination. Finally, 15 cc blood will be drawn from the heart.

SUMMARY:
Rationale In a very short time corona virus disease 2019 (COVID-19) has become a pandemic with high morbidity and mortality. The main cause of death is respiratory failure including acute respiratory distress syndrome, however the exact mechanisms and other underlying pathology is currently not yet known. In the current setting of the COVID-19 pandemic complete autopsies seem too risky due to the risk of SARS CoV-2 transmission. Yet, as so little is known, additional histopathological, microbiological and virologic study of tissue of deceased COVID-19 patients will provide important clinical and pathophysiological information. Minimal invasive autopsy combined with postmortem imaging seems therefore an optimal method combining safety on the one hand yet proving significant information on the other.

This study aims to determine the cause of death and attributable conditions in deceased COVID-19 patients. This will be performed using post-mortem CT-scanning plus CT-guided MIA to obtain tissue for further histological, microbiological and pathological diagnostics. In addition, the pathophysiology of COVID-19 will be examined by further tissue analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with COVID-19 that die during hospitalization in Jessa hospital. COVID-19 is defined as either a positive SARS CoV-2 PCR result OR a high clinical suspicion combined with typical radiologic findings in the absence of an alternative explanation for the clinical picture.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Determination of cause of death and contributing factors based on clinical, radiological, microbiological and histopathological data of the deceased patient | up to one month
  For each individual patient the cause of death and contributing factors will be assessed. For each individual these diagnoses will be made during a meeting of a multidisciplinary team consisting of at least an infectious diseases physician, a radiologist and a pathologist. On a case to case basis, additional medical specialists can be asked to attend, including an intensive care specialist, a geriatrician and/or a microbiologist.
  During the meetings, the clinical, radiological, microbiological and histopathological data will be presented to all attending specialists. The final diagnoses will be based on consensus.
  Outcomes will be reported as proportions with a 95% confidence interval.

SECONDARY OUTCOMES:
Detailed description of the postmortem radiological changes induced by COVID-19 | up to one month
  The radiological findings will be systematically scored as absent or present. These findings will be reported as proportions with a 95% confidence interval.
Detailed description of the postmortem histopathological changes induced by COVID-19 | up to one month
  On the basis of clinical observations at this moment in time correlations will be done between the renal histology findings of the patients with and without renal failure at death as well as between the cardiac histology findings of the patients with and without clinical signs of myocarditis. However, in the light of continuous clinical observations and new insights, this may be expanded in the future. Outcomes will be reported as proportions with a 95% confidence interval.
Postmortem quantity of viral RNA | up to one month
  Describe the quantity of viral RNA in the different tissues and relate this to the clinical, radiological and histopathological findings.
Postmortem disease mechanisms at cellular level | up to one month
  Study in detail the disease mechanisms at cellular level (including ACE-2 receptor expression in relation to quantity of viral RNA) in the different tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Janneke Cox, MD, PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Belgium

REFERENCES:
- [Derived] Van Cleemput J, van Snippenberg W, Lambrechts L, Dendooven A, D'Onofrio V, Couck L, Trypsteen W, Vanrusselt J, Theuns S, Vereecke N, van den Bosch TPP, Lammens M, Driessen A, Achten R, Bracke KR, Van den Broeck W, Von der Thusen J, Nauwynck H, Van Dorpe J, Gerlo S, Maes P, Cox J, Vandekerckhove L. Organ-specific genome diversity of replication-competent SARS-CoV-2. Nat Commun. 2021 Nov 16;12(1):6612. doi: 10.1038/s41467-021-26884-7. PMID 34785663
- [Derived] D'Onofrio V, Donders E, Vanden Abeele ME, Dubois J, Cartuyvels R, Achten R, Lammens M, Dendooven A, Driessen A, Augsburg L, Vanrusselt J, Cox J. The clinical value of minimal invasive autopsy in COVID-19 patients. PLoS One. 2020 Nov 11;15(11):e0242300. doi: 10.1371/journal.pone.0242300. eCollection 2020. PMID 33175911